CLINICAL TRIAL: NCT01676038
Title: Radiographic Analysis Comparing Pinless-Navigated and Conventional Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Pinless-Navigated Versus Conventional Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011/519/D
Record Dates: First submitted 2012-08-03; First posted 2012-08-30 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Arthropathy of Knee
Keywords: Total Knee Replacement, Computer-Assisted Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pinless-Navigated Total Knee Arthroplasty (Active Comparator): The patients underwent total knee arthroplasty using a Pinless-Navigated system that is designed to restore the mechanical alignment of the lower limb.
  Interventions: Procedure: Pinless-Navigated Total Knee Arthroplasty
- Conventional Total Knee Arthroplasty (Active Comparator): The patients underwent total knee arthroplasty using conventional technique.
  Interventions: Procedure: Conventional Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Pinless-Navigated Total Knee Arthroplasty — Brainlab VectorVision Knee 2.5 Navigation System
  Arms: Pinless-Navigated Total Knee Arthroplasty
Procedure: Conventional Total Knee Arthroplasty — Conventional technique.
  Arms: Conventional Total Knee Arthroplasty

SUMMARY:
The success of total knee arthroplasty depends on a number of factors including pre-operative range of movement, obesity, medical comorbidities, prosthesis design, preparation and implantation of the prosthesis, soft tissue balancing, as well as implants alignment. Optimal placement of the implants within 3° of the mechanical axis of the lower limb has been proven to reduce wear and early implant failure.

Compared to conventional techniques, computer-Aided Navigation total knee arthroplasty has been widely used in the last decade and have been proven to improve the accuracy of prosthesis placement and lower limb alignment by reducing the number of outliers with more than 3° deviation from the mechanical axis. However, its use also involves a steep learning curve, high initial capital cost and longer duration of surgery.

Traditional computer-navigated TKA using optical tracking systems also requires fixation of the femoral and tibial reference arrays to bone using anchoring pins. Complications reported with the use of these pins include either femoral or tibial fracture, pin site pain, pin site infection and osteomyelitis. The investigators study aims to investigate the accuracy of a new pinless navigation system for TKA that will avoid these complications.

DETAILED DESCRIPTION:
The duration of surgery and length of hospital stay were recorded for all patients. Three radiographic measurements were recorded on the coronal films: 1) Hip-Knee-Ankle Angle (HKA), the angle formed by the mechanical axis of the femur (line between the centre of the femoral head and the centre of the knee) and the mechanical axis of the tibia (line between the centre of the talus and the centre of the knee); 2) Coronal Femoral-Component Angle (CFA), the angle formed by the femoral component and the mechanical axis of the femur; 3) Coronal Tibia-Component Angle (CTA), the angle formed by the tibia base plate and the mechanical axis of the tibia. The post-operative radiographic measurements were compared with the intra-operative readings from the pinless navigation system. The accepted values used in our study for normal alignment were: 1) 0° ± 3° varus/valgus for HKA; 2) perpendicular (± 3°) to the mechanical axis of the femur; 3) perpendicular (± 3°) to the mechanical axis of the tibia.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 45 and 90 diagnosed with osteoarthritis of the knee and scheduled for unilateral total knee replacement.

Exclusion Criteria:

* Patients coming for revision total knee arthroplasty
* Patients diagnosed with inflammatory arthritis

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Radiographic analysis | Up till 1 year
  The number of outliers and mean value of: 1) Hip-Knee-Ankle Angle (HKA), the angle formed by the mechanical axis of the femur (line between the centre of the femoral head and the centre of the knee) and the mechanical axis of the tibia (line between the centre of the talus and the centre of the knee); 2) Coronal Femoral-Component Angle (CFA), the angle formed by the femoral component and the mechanical axis of the femur; 3) Coronal Tibia-Component Angle (CTA), the angle formed by the tibia base plate and the mechanical axis of the tibia.

SECONDARY OUTCOMES:
Duration of surgery | Up till 1 year
  Comparing the mean duration of surgery for both surgical arms.

CONTACTS AND LOCATIONS:
Overall Officials: Pak Lin Chin, FRCS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore